CLINICAL TRIAL: NCT07202754
Title: The Impact of Procedural Complications on Long-Term Mortality in Complex Coronary Interventions: The Multicenter COMPLEX-ANATOLIA Study
Brief Title: Procedural Complications and Long-Term Mortality in Complex Coronary Interventions
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Mehmet Akif Ersoy Educational and Training Hospital (Other Government)
Collaborators: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government); Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other); Istanbul Training and Research Hospital (Other Government); Sisli Hamidiye Etfal Training and Research Hospital (Other); Bagcilar Training and Research Hospital (Other Government); Ankara Etlik City Hospital (Other Government); Ankara Bilkent Sehir Hastanesi (Other); Bursa Yuksek Ihtisas Training and Research Hospital (Other Government); Bursa City Hospital (Other Government); Ege University (Other); Kocaeli University (Other); Trakya University (Other); Van Training and Research Hospital (Other Government); Cigli Regional Training Hospital (Other); Istanbul University - Cerrahpasa (Other); University of Yalova (Other)
Responsible Party: Principal Investigator, Ahmet Guner, Principal Investigator, Istanbul Mehmet Akif Ersoy Educational and Training Hospital
Other Study IDs: 2025.04-35
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Complex Coronary Artery Disease
Keywords: Complications, death, major adverse cardiac events, target vessel revascularization
MeSH Terms: conditions — Death; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Non-fatal complications (+)
- Group 2: Non-fatal complications (-)

SUMMARY:
The relative risks for different non-fatal intraprocedural complications during complex percutaneous coronary intervention (PCI) on subsequent mortality have not been described. This study aimed to assess the association between non-fatal intraprocedural complications and late mortality after complex coronary PCI.

DETAILED DESCRIPTION:
Complex coronary lesions include chronic total occlusion, osteal epicardial lesions, long (diffuse) coronary disease, severe calcific lesions, true bifurcation disease, left main coronary lesion, lesions with severe thrombus, and in-stent restenosis. Non-fatal intraprocedural complications included abrupt occlusion, worsening of thrombolysis in myocardial infarction (TIMI) flow grade (TIMI < 3), major dissection (greater than type B), occurrence of thrombus formation, perforation of the main vessel or side branch, malignant arrhythmias, stroke/transient ischemic attack, and non-coronary major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex coronary disease
* Aged 18-85 years

Exclusion Criteria:

* Patients diagnosed with cardiogenic shock
* Coronary lesions with non-complex features
* Percutaneous coronary intervention with a bare metal stent
* Patient life expectancy <1 year
* Known relevant allergies
* Absence of all medical records
* Patients with early discontinuation of dual antiplatelet therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Complex coronary lesions include chronic total occlusion, osteal epicardial lesions, long (diffuse) coronary disease, severe calcific lesions, true bifurcation disease, left main coronary lesion, lesions with severe thrombus, and in-stent restenosis.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Death | up to 60 months
  All cause death

IPD SHARING:
Plan to Share IPD: No